CLINICAL TRIAL: NCT04822207
Title: Effect of Acupuncture on the Clinical Outcome of IVF-ET in Patients With Recurrent Implantation Failure: a Multicenter Randomized Controlled Trial
Brief Title: Effect of Acupuncture on the Clinical Outcome of IVF-ET in Patients With Recurrent Implantation Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ShangHai Ji Ai Genetics & IVF Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JIAI 2021-01
Record Dates: First submitted 2021-03-25; First posted 2021-03-30 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-03

CONDITIONS: Acupuncture; Recurrent Implantation Failure
Keywords: acupuncture; recurrent implantation failure
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture group (Experimental): In the acupuncture group, those patients undergo acupuncture at the beginning of embryo transfer cycle three times a week until 14 days after embryo transfer. These patients should be checked including endometrial receptivity index and fill in SAS anxiety scale form.
  Interventions: Procedure: acupuncture
- Control group (No Intervention): In the control group, these patients do not receive any treatments during embryo transfer cycle. These patients should be checked including endometrial receptivity index and fill in SAS anxiety scale form.

INTERVENTIONS:
Procedure: acupuncture — Patients undergo acupuncture at the beginning of embryo transfer cycle three times a week until 14 days after embryo transfer. Every acupuncture lasts 20 minutes.
  Arms: Acupuncture group

SUMMARY:
In order to explore the effect of acupuncture on the clinical outcome of IVF-ET in patients with recurrent implantation failure, the patients divide into the experimental group or the control group. In the experimental group, those patients undergo acupuncture at the beginning of embryo transfer cycle three times a week until 14 days after embryo transfer. In the control group, those patients do not receive any treatments during embryo transfer cycle. Statistical analysis of the two groups of primary endpoint and secondary endpoint are done.

DETAILED DESCRIPTION:
In the field of assisted reproduction techonology, there are still 10% of patients with recurrent implantation failure. In order to explore the effect of acupuncture on the clinical outcome of IVF-ET in patients with recurrent implantation failure, the patients divide into the experimental group or the control group. In the experimental group, those patients undergo acupuncture at the beginning of embryo transfer cycle three times a week until 14 days after embryo transfer. In the control group, those patients do not receive any treatments during embryo transfer cycle. Both of two group patients are checked including endometrial receptivity index and fill in SAS anxiety scale form. Statistical analysis of the two groups of primary endpoint (clinical pregnancy rate) and secondary endpoint (embryo implantation rate, biochemical pregnancy rate, early pregnancy loss rate, ongoing pregnancy rate, live birth rate)are done.

ELIGIBILITY:
Inclusion Criteria:

1. A: ≥ 3 times embryo transfer failures，and at least accumulated 4 high-quality embryos were transferred

B: Two times consecutive embryo transfers failures, at least accumulated 4 high-quality embryos were transferred

2. Undergo IVF / ICSI / PGT;

3. Transfer 1-2 D3 cleavage embryos or blastocysts in IVF / ICSI and transfer 1 blastocyst in PGT;

4. 20-38 years old female

5. Sign the informed consent voluntarily.

Exclusion Criteria:

1. Contraindications for pregnancy or assisted reproductive technology;
2. Chromosome abnormality of husband or wife (except polymorphism);
3. Abnormal gene diseases;
4. Untreated of uterine diseases that affect the uterine cavity morphology (uterine malformation, submucous myoma, adenomyosis, endometriosis and endometriosis etc.);
5. AMH < 1.1ng/ml or AFC < 7;
6. The most thickness of endometrium is less than 7 millimeter;
7. Those who have more than 2 times clinical pregnancy abortion;
8. Patients with serious primary diseases including cardiovascular, cerebrovascular, liver, kidney and hematopoietic system and mental diseases
9. The treatment (such as acupuncture and traditional Chinese Medicine) related to help pregnancy had been carried out in the last 3 months.

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 310 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 6 months
  Clinical pregnancy will be defined as ultrasonographic evidence of an intrauterine sac with or without a fetal heart at the 6th gestational week.

SECONDARY OUTCOMES:
embryo implantation rate | 6 months
  The embryo implantation rate (IR) will be calculated as the number of gestational sacs per embryo transferred
biochemical pregnancy rate | 6 months
  Biochemical pregnancy will be defined by a serum HCG level ≥5.0 mIU/ml approximately 14 days after embryo transfer
early pregnancy loss rate | 6 months
  Early pregnancy loss will be considered pregnancy loss occurring after detection of a clinical pregnancy up to the 12th week of pregnancy
ongoing pregnancy rate | 6 months
  OPR was calculated by considering all viable intrauterine pregnancy progressing beyond 12 weeks of gestation.
live birth rate | 12 mongths
  Live birth rates were calculated based on the total number of live births > 20 weeks' gestation over the total number of ongoing pregnancies.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxi Sun, Study Chair — Obstetrics and Gynecology Hospital affiliated to Fudan University
Locations (1):
- Shanghai Ji Ai Genetics & IVF Institute, Obstetrics and Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Westergaard LG, Mao Q, Krogslund M, Sandrini S, Lenz S, Grinsted J. Acupuncture on the day of embryo transfer significantly improves the reproductive outcome in infertile women: a prospective, randomized trial. Fertil Steril. 2006 May;85(5):1341-6. doi: 10.1016/j.fertnstert.2005.08.070. Epub 2006 Apr 5. PMID 16600232
- [Background] Paulus WE, Zhang M, Strehler E, El-Danasouri I, Sterzik K. Influence of acupuncture on the pregnancy rate in patients who undergo assisted reproduction therapy. Fertil Steril. 2002 Apr;77(4):721-4. doi: 10.1016/s0015-0282(01)03273-3. PMID 11937123
- [Background] Dieterle S, Ying G, Hatzmann W, Neuer A. Effect of acupuncture on the outcome of in vitro fertilization and intracytoplasmic sperm injection: a randomized, prospective, controlled clinical study. Fertil Steril. 2006 May;85(5):1347-51. doi: 10.1016/j.fertnstert.2005.09.062. Epub 2006 Apr 17. PMID 16616748